CLINICAL TRIAL: NCT03343223
Title: A Brief, Pragmatic Experiment to Determine the Impact of a Public-health-partnered Tele-pharmacist Model for PrEP Delivery in a Rural State
Brief Title: Rural PrEP Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Ohl (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Michael Ohl, Associate Professor of Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201711710
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1. Public health personnel identify PrEP-eligible clients.
  2. PrEP-eligible clients are given a list of PrEP providers in Iowa and a brochure with info on getting PrEP. Clients are referred to a PrEP navigator, who facilitates linkage to clients' choice of TelePrEP or to community PreP providers.
  3. Public health clients choosing TelePrEP complete a video visit with the tele-pharmacist and obtain PrEP relevant lab tests.
  4. PrEP medication is mailed to the client and follow up video visits and lab testing are performed.
  5. Within 7 days of enrollment, the subject will complete a survey regarding PrEP beliefs (20 minutes).
  6. 30 to 40 days after enrollment, the subject will complete a second survey with 4 questions about initiation of PrEP since study enrollment (10 minutes).
  7. 6 months following enrollment, a study team member will obtain medical records for the subject from PrEP providers in Iowa to determine if the subject has initiated and been retained in PrEP.
  Interventions: Behavioral: Intervention Group
- Control Group (No Intervention): 1. Public health personnel identify PrEP-eligible.
  2. Public health personnel give PrEP-eligible clients a list of PrEP providers in Iowa, and a brochure with information on getting PrEP.
  3. The client initiates contact with a PrEP provider in Iowa and schedules an appointment.
  4. PrEP medication is mailed to the client and follow up video visits and lab testing are performed.
  5. Within 7 days of enrollment, the subject will complete a survey regarding PrEP beliefs (20 minutes).
  6. 30 to 40 days after enrollment, the subject will complete a second survey with 4 questions about initiation of PrEP since study enrollment (10 minutes).
  7. 6 months following enrollment, a study team member will obtain medical records for the subject from PrEP providers in Iowa to determine if the subject has initiated and been retained in PrEP.

INTERVENTIONS:
Behavioral: Intervention Group — The goal of this research study is to evaluate the preliminary impact of a public-health-partnered tele-pharmacist model for pre-exposure prophylaxis (PrEP) delivery in a rural state ("TelePrEP"). In brief, PrEP involves daily use of a medication (i.e. Truvada) to prevent HIV infection among people at risk for infection due to sexual exposure or needle sharing.
  Arms: Intervention Group

SUMMARY:
The goal of this research study is to evaluate the preliminary impact of a public-health-partnered tele-pharmacist model for pre-exposure prophylaxis (PrEP) delivery in a rural state ("TelePrEP"). In brief, PrEP involves daily use of a medication (i.e. Truvada) to prevent HIV infection among people at risk for infection due to sexual exposure or needle sharing. In this study, PrEP eligible rural and small urban-dwelling public health clients wil be enrolled in a prospective study to follow their progression through PrEP care following public health referrals. The study will involve a baseline survey to gather data on participant beliefs and attitudes about PrEP and a follow up telephone survey 30-40 days later to ascertain whether participants have engaged in PrEP. Medical records will be requested as a second method to determine whether participants have started PrEP and whether they are still using PrEP after six months. The hypotheses that PrEP initiation and retention are higher in regions with TelePrEP programs will be tested against control regions.

DETAILED DESCRIPTION:
The Iowa Department of Public Health (IDPH) and The University of Iowa (UI) have collaborated to develop a public-health-partnered tele-pharmacist model that meets these needs ("TelePrEP"). TelePrEP was developed and piloted as a quality improvement program and uses only standard of care interventions (e.g. PrEP) and routinely applied healthcare delivery strategies (e.g. telemedicine, pharmacist collaborative practice models). In overview, TelePrEP begins by systematically identifying clients with PrEP indications in county public health clinics and affiliated sexually-transmitted disease (STD) programs serving rural and small urban communities in Iowa. Public health personnel then refer clients with PrEP indications to a tele-pharmacist service at UIHC that uses mobile video visits, locally-obtained laboratory studies, and medication delivery by mail to provide PrEP, without requiring in-person provider visits. The overall goal is to improve PrEP access and engagement in rural and small urban areas by systematically identifying high risk-individuals in public health programs, and referring these individuals to a geographically-scalable tele-pharmacist PrEP clinic that overcomes barriers related to distance and stigma.

The TelePrEP program was piloted locally in Johnson County, and in 2018 the IDPH and UI will collaborate to scale it up across Iowa. In parallel with scale up of the TelePrEP program, a research study will be conducted to determine the impact of TelePrEP on PrEP use among rural and small urban -dwelling public health clients. In a quasi-experimental study, the local public health departments in Iowa and their affiliated HIV/STD programs will be divided into TelePrEP intervention and control groups, based on geographic region. This is appropriate because it will not be feasible to implement the TelePrEP program in all Public health sites simultaneously, so some sites will start the program later than others by necessity. Public health personnel in control regions will refer PrEP-eligible clients to available community-based PrEP providers, the current "standard of care." Public health personnel in TelePrEP intervention regions will refer clients to their choice of in-person visits with available community PrEP providers or TelePrEP.

Primary Objective: Estimate the impact of TelePrEP on the overall rate of PrEP engagement among rural and small urban public health clients.

* To compare total rates of PrEP engagement among PrEP-eligible clients in intervention and control regions, defining PrEP engagement as any provider visit (i.e. in-person community provider visit or tele-pharmacist) to discuss PrEP AND a Truvada® prescription within 30 days of public health referral.
* Hypothesis 1: TelePrEP will increase PrEP engagement from 5% in control regions to 25% in TelePrEP intervention regions.

Secondary Objective: Quantify retention of public health clients in TelePrEP.

* Following PrEP engagement, we will measure the proportion of clients who are retained in PrEP six months following engagement, defining retention as a tele-pharmacist video or community PrEP provider visit between days 150 and 210 with self-reported Truvada® use in the past week.
* Hypothesis 2a: Over 50% of clients engaging in TelePrEP will be retained at 6 months.
* Hypothesis 2b: Retention in PrEP will be greater in TelePrEP regions.

ELIGIBILITY:
Inclusion Criteria:

1. Public health client in CTR-PS programs
2. Rural or small urban-dwelling residents (Iowa residence NOT residing in Polk, Linn, Scott, or Pottawattamie counties)
3. Adults (age 18+)
4. Referred by public health for PrEP based on:

HIV-negative by recent (< or = 14 days) testing AND one of following

1. men sexually active with male partner(s) in the past six months, not in a monogamous partnership with a recently-tested HIV negative man, and reporting either anal sex without condoms in the past six months, any STI in past six months, or relationship with an HIV-positive partner,

   OR
2. sexually-active heterosexual men and women not in a monogamous relationship with an HIV-negative partner and reporting either condom-less sex with partners of unknown HIV status at high risk for HIV infection, or an ongoing sexual relationship with an HIV-positive partner,

   OR
3. intravenous drug users (IDU) injecting drugs in the past six months and reporting either sharing of drug equipment, receipt of methadone or buprenorphine treatment in the past six months, or risk of sexual acquisition.

Exclusion Criteria:

1. Self-reported current PrEP use
2. Self-reported inability to access a computer, smartphone, or tablet.
3. Residence in a large urban County (i.e. Polk, Linn, Scott, Pottawattamie)
4. HIV positive status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Impact of TelePrEP on overall rate of PrEP engagement | 30 days
  Rates of PrEP engagement among PrEP-eligible clients in intervention and control regions

SECONDARY OUTCOMES:
Retention of clients in TelePrEP | 6 months
  Proportion of clients who are retained in PrEP six months following engagement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No